CLINICAL TRIAL: NCT04349306
Title: An Open-label, Single-arm, Multi-center Study to Evaluate the Efficacy and Safety of Rasburicase (Fasturtec) in the Prevention and Treatment of Hyperuricemia in Pediatric Patients With Non-Hodgkin¿s Lymphoma and Acute Leukemia
Brief Title: Evaluate the Efficacy and Safety of Rasburicase (Fasturtec®) in the Prevention and Treatment of Hyperuricemia in Pediatric Patients With Non-Hodgkin's Lymphoma and Acute Leukemia
Acronym: RAISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RASBUL09107; U1111-1233-0737 (Other: UTN)
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rasburicase (Experimental): rasburicase 0.20 mg/kg/day by intravenous (IV) over 30 minutes for 1 to 5 days according to the level of plasma uric acid or Investigator's clinical judgement
  Interventions: Drug: RASBURICASE SR29142

INTERVENTIONS:
Drug: RASBURICASE SR29142 — Pharmaceutical form:solution for infusion Route of administration: intravenous

SUMMARY:
Primary Objective:

To evaluate safety of rasburicase in pediatric patients with NHL and AL

Secondary Objective:

To assess efficacy of rasburicase for prevention and treatment of hyperuricemia

DETAILED DESCRIPTION:
Study duration per participants is approximatively 14 days including a 5-day treatment period.

ELIGIBILITY:
Inclusion criteria :

* Patient or parent/legal guardian is willing and able to provide signed informed consent, and if required, the patient is willing to provide assent.
* Children or adolescent aged 2 to 18 years old (inclusive) at time of signing of informed consent.
* At screening, the patient is expected to have a minimum life expectancy of 45 days and has a performance status (PS) no greater than 3 on the Eastern Cooperative Oncology Group (ECOG) scale, or a PS no less than 30 on the Lansky score as per the Investigator's preference (see Appendix D for ECOG and Lansky scale).
* Newly diagnosed NHL or AL who is at the initiation of or during the first cycle of chemotherapy,baseline blood uric acid greater than 8 mg/dL (473 mol/L) at screening.
* If newly diagnosed NHL patient with blood uric acid no greater than 8 mg/dL at screening, the patient must be diagnosed with Stage III or IV non-Hodgkin's lymphoma with high tumor burden which will be high risk of TLS defined, with one or more of following below: A. Burkitt lymphoma/leukemia or -lymphoblastic lymphoma, and/or B. Has at least one of lymph node or tumor, the diameter >5 cm, and/or C. Lactate dehydrogenase (LDH) no less than 2 times the upper limit of normal (ULN).
* If newly diagnosed AL patient is with blood uric acid no greater than 8 mg/dL at the screening but with a high risk of TLS defined with one of the following below criteria: A. White blood cell (WBC) no less than 100.0 10-9/L, or B. WBC < 100.0 10-9/L with LDH no less than 2 ULN.
* The patient will receive the chemotherapy, and will be confined in hospital for at least 14 days after first dose of rasburicase.

Exclusion criteria:

* Acute promyelocytic leukemia
* Patient who has been treated or planned to receive allopurinol within 72 hours of rasburicase administration.
* Patients with abnormal liver or renal function: alanine aminotransferase (ALT) >5 ULN, total bilirubin >3 ULN, serum creatinine >3 ULN.
* Documented history of hereditary allergy or asthma.
* Patients with known deficiency of glucose-6-phosphate dehydrogenase (G6PD), or a history of hemolytic disease or methemoglobinemia.
* Patients with severe infection or active bleeding.
* Previous therapy with urate oxidase.
* Hypersensitive reaction against rasburicase or any of the other ingredients of the study drug.
* Patient is not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or patients potentially at risk of noncompliance to study procedures.
* Pregnant or breastfeeding woman.
* Woman of childbearing potential (WOCBP) not protected by highly-effective method(s) of birth control and/or who are unwilling or unable to be tested for pregnancy (see contraceptive guidance in Appendix A).
* Male participant with a female partner of childbearing potential not protected by highly-effective method(s) of birth control

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs | Day 1 to Day 7
  Incidence of AE or SAE will be summarized as the number and percentage of subjects who experienced any AE or SAE during the treatment period.

SECONDARY OUTCOMES:
Number of responders after completion of rasburicase treatment under chemotherapy | Day 1 to Day 7
  Response will be defined as achievement of normal uric acid levels (≤ 8.0 mg/dL) in those patients whose uric acid levels are >8.0 mg/dL.
Proportion of patients who can maintain the normal uric acid levels throughout the study | Day 1 to Day 7
  In those patients whose baseline plasma uric acid levels are ≤ 8 mg/dL but with a high risk of TLS.
Percentage of the maximum decreasing degree of plasma uric acid level from baseline | Day 1 to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- investigational site CHINA, China, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org